CLINICAL TRIAL: NCT06816849
Title: The Role of Hydration in the Management of Pediatric Primary Headaches: A Pilot Study
Brief Title: Hydration in Children and Adolescents With Primary Headaches
Acronym: H20KIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KME:0120-423/2023-2711-6; Master Research (Other: University Medical Centre Ljubljana and University of Ljubljana, Slovenia)
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-03

CONDITIONS: Primary Headaches (Includes Migraines, Tension, Cluster Headaches); Hydration; Adolescent; Children
Keywords: primary headache; pediatric; children; hydration; water intake
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recommended fluid intake (Experimental): All participants received personalized consultation from a dietitian on adequate fluid intake and the selection of drinks based on dietary guidelines. They were required to follow the intervention for four months.
  Interventions: Other: Recommended water intake

INTERVENTIONS:
Other: Recommended water intake — All participants received personalized consultation from a dietitian on adequate fluid intake and the selection of drinks based on dietary guidelines. They were required to follow the intervention for four months.

SUMMARY:
The aim of this study is to investigate the role of hydration and fluid intake in children and adolescents with primary headaches.

DETAILED DESCRIPTION:
Headches are one of the key factors affecting or even limiting the health and well-being of children and adolescents. Lifestyle recommendations could help reduce the risk of chronic headaches and improve overall well-being in this population. In clinical practice, adequate fluid intake is one of the general recommendations for headache management. However, scientific literature on the role of hydration and fluid intake in headaches is limited. To date, all studies have been conducted on adults, and no studies have examined this topic in the pediatric population.

As the first interventional study investigating the impact of adequate fluid intake on headaches in children and adolescents, our study will make a significant contribution to understanding the role of hydration in headache management and developing recommendations for improving headache control in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years.
* Able to provide informed consent and willing to complete follow-up visits.
* Primary headaches.
* At least 1 headache per month.
* Presence of headaches for at least 3 months or longer.

Exclusion Criteria:

* Secondary headaches.
* Without headaches for 3 months or more.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Headache frequency | 4 months
  Number of headache episodes over last three months.
Headache intensity | 4 months
  Headache severity measured with the Visual Analog Scale (0 - 10).
Headache duration | 4 months
  Average length of headache episode measured in minutes.

SECONDARY OUTCOMES:
Change in total body water | 4 months
  Change in total body water (liter and %) assessed with bioelectrical impedance analysis (BIA 101 AKern) following the intervention.
Effect of nutritional advice on type of drink they have choosen | 4 months
  Type of fluid they had increased during intervention.
Change in extracellular water | 4 months
  Change in extracellular water (liter and %) assessed with bioelectrical impedance analysis (BIA 101 AKern) following the intervention.
Change in phase angle | 4 months
  Change in phase angle (°) assessed with bioelectrical impedance analysis (BIA 101 AKern) following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spigt MG, Kuijper EC, Schayck CP, Troost J, Knipschild PG, Linssen VM, Knottnerus JA. Increasing the daily water intake for the prophylactic treatment of headache: a pilot trial. Eur J Neurol. 2005 Sep;12(9):715-8. doi: 10.1111/j.1468-1331.2005.01081.x. PMID 16128874
- [Result] Spigt M, Weerkamp N, Troost J, van Schayck CP, Knottnerus JA. A randomized trial on the effects of regular water intake in patients with recurrent headaches. Fam Pract. 2012 Aug;29(4):370-5. doi: 10.1093/fampra/cmr112. Epub 2011 Nov 23. PMID 22113647
- [Result] Khorsha F, Mirzababaei A, Togha M, Mirzaei K. Association of drinking water and migraine headache severity. J Clin Neurosci. 2020 Jul;77:81-84. doi: 10.1016/j.jocn.2020.05.034. Epub 2020 May 20. PMID 32446809